CLINICAL TRIAL: NCT07295080
Title: Comparison of Dural Puncture Epidural and Standard Epidural Anesthesia Techniques in Elective Cesarean Deliveries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Esra Uyar Türkyılmaz, associate professor,MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1251153
Record Dates: First submitted 2025-11-20; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Regional Anaesthesia in Cesarean Operations
Keywords: dural puncture epidural anesthesia; epidural anesthesia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dural puncture epidural (Experimental): The epidural space will be accessed using an 18G epidural needle, followed by dural puncture with a 27G spinal needle. Without administering any drug into the cerebrospinal fluid (CSF), an epidural catheter will then be inserted, through which anesthesia will be administered.Its placement will be confirmed with a test dose of 2 ml of 2% lidocaine. Following the test dose (after excluding signs of intrathecal or intravenous injection), a mixture consisting of 7.5 ml of 2% prilocaine, 7.5 ml of 0.5% bupivacaine, and 100 µg of fentanyl (2 ml) will be administered in 5-ml increments at 3-minute intervals. At the completion of the injection (t0), the patient will be placed in the supine position with a 10-degree left tilt. Sensory block level will be assessed every minute using the pinprick test. Bilateral sensory block at the T5 dermatome will be accepted as adequate surgical anaesthesia.
  Interventions: Other: Dural puncture epidural (DPE) anaesthesia
- standart epidural anesthesia (Active Comparator): The epidural space will be accessed using an 18G epidural needle. An epidural catheter will then be inserted, through which anesthesia will be administered.Its placement will be confirmed with a test dose of 2 ml of 2% lidocaine. Following the test dose (after excluding signs of intrathecal or intravenous injection), a mixture consisting of 7.5 ml of 2% prilocaine, 7.5 ml of 0.5% bupivacaine, and 100 µg of fentanyl (2 ml) will be administered in 5-ml increments at 3-minute intervals. At the completion of the injection (t0), the patient will be placed in the supine position with a 10-degree left tilt. Sensory block level will be assessed every minute using the pinprick test. Bilateral sensory block at the T5 dermatome will be accepted as adequate surgical anaesthesia.
  Interventions: Other: standart epidural anesthesia

INTERVENTIONS:
Other: Dural puncture epidural (DPE) anaesthesia — The epidural space will be accessed using an 18G epidural needle, followed by dural puncture with a 27G spinal needle. Without administering any drug into the cerebrospinal fluid (CSF), an epidural catheter will then be inserted, through which anesthesia will be administered.Its placement will be confirmed with a test dose of 2 ml of 2% lidocaine. Following the test dose (after excluding signs of intrathecal or intravenous injection), a mixture consisting of 7.5 ml of 2% prilocaine, 7.5 ml of 0.5% bupivacaine, and 100 µg of fentanyl (2 ml) will be administered in 5-ml increments at 3-minute intervals.
  Arms: dural puncture epidural
Other: standart epidural anesthesia — The epidural space will be accessed using an 18G epidural needle. An epidural catheter will then be inserted, through which anesthesia will be administered.Its placement will be confirmed with a test dose of 2 ml of 2% lidocaine. Following the test dose (after excluding signs of intrathecal or intravenous injection), a mixture consisting of 7.5 ml of 2% prilocaine, 7.5 ml of 0.5% bupivacaine, and 100 µg of fentanyl (2 ml) will be administered in 5-ml increments at 3-minute intervals.
  Arms: standart epidural anesthesia

SUMMARY:
Neuraxial techniques are the most effective form of labor analgesia in contemporary obstetric anesthesia practice, predominantly through the use of epidural (EPL) and combined spinal-epidural (CSE) techniques. Although drug combinations employed in these methods have advanced, the onset time, block quality, and side effect profiles of both techniques still require further improvement.

The epidural technique is associated with minimal side effects; however, it may occasionally present variable block characteristics such as slow onset, inadequate sacral spread, unilateral or patchy sensory block, motor impairment, and epidural catheter failure.

The dural puncture epidural (DPE) technique is performed by inserting a spinal needle through the shaft of the epidural needle to create a single dural perforation, after which an epidural catheter is placed into the epidural space without administering any drugs into the cerebrospinal fluid (CSF). All medications for analgesia or anesthesia are delivered into the epidural space via the catheter. The dural puncture is thought to provide a conduit that facilitates the translocation of drugs from the epidural space into the subarachnoid space, which is believed to account for the clinical features observed with the dural puncture epidural technique advantageous in obstetric patients. Additionally, the process of dural puncture with a spinal needle through the epidural needle allows cerebrospinal fluid return to serve as a "confirmatory" definitive endpoint for the position of the epidural needle tip within the epidural space.

The investigators designed this study to determine whether the dural puncture epidural technique, compared with epidural, could improve the onset time and block characteristics of anesthesia in elective cesarean deliveries.

Compared with the epidural technique, the dural puncture epidural approach has been shown to improve the onset of sacral block as well as the spread of anesthesia and analgesia-characteristics that are particularly advantageous in obstetric patients. Additionally, the process of dural puncture with a spinal needle through the epidural needle allows cerebrospinal fluid return to serve as a "confirmatory" definitive endpoint for the position of the epidural needle tip within the epidural space.

The investigators designed this study to determine whether the dural puncture epidural technique, compared with epidural, could improve the onset time and block characteristics of anesthesia in elective cesarean deliveries.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of dural puncture epidural (DPE) versus standard epidural anesthesia on the time to surgical anesthesia onset in patients scheduled for elective cesarean section.

• Study Population:

Pregnant women undergoing elective cesarean section

• Compared Techniques:

Dural Puncture Epidural Group → A dural puncture will be performed with a 27G spinal needle before the placement of the epidural catheter.

Standard Epidural Group → An epidural catheter will be placed directly without dural puncture.

• Primary Outcome:

Time from anesthesia administration to onset of surgical anesthesia (defined as time to achieve sensory block at the T5 dermatome level).

• Secondary Outcomes:

Incidence of hypotension

Intraoperative ephedrine requirement

Need for additional doses

Post-dural puncture headache (PDPH)

Time to regression of sensory block

Motor block assessment (Bromage scale)

Study Design:

Prospective: Patients will be identified before anesthesia administration and evaluated going forward.

Randomized: Patients will be randomly assigned to either the dural ponksiyon epidural or standard epidural group.

Controlled: The two groups will be compared to analyze the effects.

Single-Center: The study will be conducted at a single hospital. Inclusion Criteria

* Women scheduled for elective cesarean delivery
* No comorbidities
* Age between 18-40 years
* Body mass index (BMI) < 35 kg/m²
* Term pregnancy ≥ 37 weeks
* No contraindications to neuraxial anesthesia (e.g., coagulopathy, infection, history of prior spinal surgery, etc.)

Parameters to Be Assessed

All parameters will be assessed by the investigator both intraoperatively and postoperatively in the ward. These include:

* Sensory block level (evaluated every minute as a study-specific parameter)
* Blood pressure
* Heart rate
* Oxygen saturation
* Requirement for ephedrine
* Requirement for additional epidural doses
* Incidence of post-dural puncture headache (at 24 and 48 hours)
* Motor block assessment (using the Bromage Scale)

Note: All evaluated parameters are part of standard monitoring, with the exception that sensory block level will be specifically assessed every minute for the purposes of this study.

-

Exclusion Criteria

* Contraindications to neuraxial anesthesia
* Refusal to participate in the study

Withdrawal and Termination Criteria

* Patient's decision to withdraw from the study
* Conversion to general anesthesia
* Administration of intrathecal and/or intravenous drugs

ELIGIBILITY:
Inclusion Criteria:

* Women scheduled for elective cesarean delivery

  * No comorbidities
  * Age between 18-40 years
  * Body mass index (BMI) < 35 kg/m²
  * Term pregnancy ≥ 37 weeks
  * No contraindications to neuraxial anesthesia (e.g., coagulopathy, infection, history of prior spinal surgery, etc.)

Exclusion Criteria:

* Contraindications to neuraxial anesthesia

  * Refusal to participate in the study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — woman
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
onset time of sensory block | 20 minutes
  The time from the administration of anesthesia to the onset of surgical anesthesia (the time it takes for the sensory block to reach the Thoracic 5 (T5) dermatome).

SECONDARY OUTCOMES:
Incidence of hypotension | perioperative
  a 20% reduction from baseline blood pressure
intraoperative ephedrine requirement | perioperative
  total intraoperative ephedrine dose
requirement for supplementery dosing | perioperative
  Failure to achieve sensory block at the Torakal 5 (T5) level within 20 minutes or the occurrence of perioperative pain
Postdural puncture headache (PDPH) | day 2
  Postoperative headaches will be evaluated at the 24th and 48th hours using the Visual Analog Scale (VAS)
Time to the onset of sensory block regression | day 1
  The duration of sensory block regression from the Thoracic 5 (T5) to the Thoracic 10 (T10) and Lumbar 1 (L1) dermatomal levels
Assessment of motor block | day 1
  The degree of motor block will be assessed using the Bromage score

CONTACTS AND LOCATIONS:
Overall Officials: esra uyar turkyilmaz, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara city hospital, Ankara, çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horcajada JP, Martinez JA, Moreno-Martinez A, Mensa J, Almela M, Soriano E. [Predictive factors of the presence of bacteremia in males with urinary infection]. Med Clin (Barc). 1999 May 29;112(19):734-5. Spanish. PMID 10394571
- [Background] Tarraga P, Garcia-Olmo D, Celada A, Garcia-Molinero Mf, Divison JA, Casado C. Colorectal cancer screening through detection of fecal occult blood in a controlled health zone. Rev Esp Enferm Dig. 1999 May;91(5):335-44. English, Spanish. PMID 10362875
- [Background] Chau A, Bibbo C, Huang CC, Elterman KG, Cappiello EC, Robinson JN, Tsen LC. Dural Puncture Epidural Technique Improves Labor Analgesia Quality With Fewer Side Effects Compared With Epidural and Combined Spinal Epidural Techniques: A Randomized Clinical Trial. Anesth Analg. 2017 Feb;124(2):560-569. doi: 10.1213/ANE.0000000000001798. PMID 28067707